CLINICAL TRIAL: NCT04247516
Title: A Study Protocol for an Online Intervention to Promote School Engagement Through Gamification in Children With Cerebral Palsy
Brief Title: A Study Protocol for an Online Intervention to Promote School Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Sílvia Lopes, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SFRH/BD/118879/2016
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
Keywords: Self-Regulation; Engagement; Gamification; Executive Function
MeSH Terms: conditions — Cerebral Palsy; Self-Control

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be developed with three groups. After obtaining informed consent from parents/caregivers, participants meeting criteria will be randomly assigned to one condition. The control group (CG) will not have access to the online platform, i.e. no intervention. The intervention group 1 (IG1) will receive on a weekly basis tasks and activities on the online platform to promote SR and SE, as well as chapters of the narrative. The intervention group 2 (IG2) will receive the same tasks and materials as IG1 but embedded with Gamification Strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Control Group (No Intervention): The standard control group (CG) will not have access to the self-regulatory (SR) intervention program.
- Online-intervention group I (IGI) (Experimental): Online-intervention group will receive on a 6-week long online intervention program. The program includes:
  i) a narrative with SR competences embedded worked on a weekly basis during an online session; ii) weekly tasks/activities will be delivered to promote the SR reflected with the narrative exploration.
  Interventions: Behavioral: Online-intervention group I (IGI)
- Online-intervention group II (IGII) (Experimental): Online-intervention group will receive on a 6-week long online intervention program. The program includes:
  i) a narrative with SR competences embedded worked on a weekly basis during an online session; ii) weekly tasks/activities will be delivered to promote the SR reflected with the narrative exploration; iii) the program includes gamification strategies with the purpose of promoting engagement in participants.
  Interventions: Behavioral: Online-intervention group II (IGII)

INTERVENTIONS:
Behavioral: Online-intervention group I (IGI) — Narrative-based online intervention program to promote self-regulatory competences.
  Arms: Online-intervention group I (IGI)
Behavioral: Online-intervention group II (IGII) — Narrative-based online intervention program to promote self-regulatory competencies plus gamification strategies.
  Arms: Online-intervention group II (IGII)

SUMMARY:
Cerebral Palsy (CP) is a neurological, non-progressive, and permanent developmental disorder that mainly affects movement and posture, with a prevalence of 3 to 4 children per 1000 live births. CP's motor impairments are often accompanied by disturbances of sensation, perception, cognition, communication, and behavior. These impairments echo in the activities of daily life, as well as in the learning process. Importantly, children with CP are especially prone to display working memory and EFs deficits, as well as difficulties in self-regulation, which might help explain some of their social and learning problems.

These children have a high risk of showing learning disabilities, which may arise before the schooling years. This risk is not exclusively determined by cognitive impairment, with children with a normative cognitive level still presenting specific learning difficulties (e.g., mathematics, reading).

Due to their clinical picture, children with disabilities, including CP, struggle with their difficulties in school. Consequently, they are prone to develop a poor School Engagement (SE) - multidimensional and multifaceted construct involving three interrelated dimensions: students' behaviors, emotions, and cognition.

In children with disabilities, one of the factors that contributes to lower SE is their high level of school absenteeism. These children miss, on average, 3 weeks of school in a school year due to health issues, which may hinder their academic performance. The promotion of SE in children with disabilities is, therefore, a priority.

To promote SE, Gamification strategies can be used. Gamification is the use of game elements (e.g., points, rewards, feedback) in non-game contexts. The potential of using Gamification is high and constitutes a unique opportunity to engage participants in specific activities, such as in intervention or learning contexts.

Therefore, through game mechanics, Gamification can be used as a tool to promote SE. This is because, it offers an attractive learning environment and converts difficult tasks into more appealing ones, motivating individuals to perform. Moreover, it enhances the degree and depth of participant engagement, rises behavior and lifestyle changes, promotes learning opportunities, motivates students, and improves intervention appeal, especially for youngsters. To conclude, this project aims to increase SE through Gamification in children with CP.

Literature has highlighted the need to focus interventions on SE and self-regulated learning (SRL) on a specific domain. Because children with CP are at high risk of presenting learning difficulties, especially in mathematics, this project will focus on mathematics performance. Moreover, SE is multidimensional, including behaviors, emotions, and cognitions related to school. Specifically, behavioral SE can be conceptualized in three levels: 1) school attendance and fulfillment of school work, 2) participation in class, and 3) active participation (e.g., doing extra school-work). Emotional SE refers to students' affective reactions and sense of connectedness with school. Finally, cognitive SE is related to personal investment in academic tasks, self-regulation, and value of the learning process. Because SRL may be compromised in children with CP, mainly due to difficulties in planning and setting goals, this project will promote SE in mathematics by developing SRL strategies in these children. SRL processes are key for students to attain their self-set goals and include competences of planning, execution, evaluation, and monitoring of the learning process. SE and SRL will be promoted through Gamification strategies on the Canvas platform.

Thus, the main purpose is to assess an intervention program with children with CP to increase SE, and enhance SRL, through Gamification Strategies in mathematics. Specifics aims:

* Embed Gamification Strategies (e.g., rewards, collaboration, competition) in the Canvas Platform using the tools already available (e.g., forum/chat);
* Develop and assess the efficacy and impact of the intervention in promoting SE, and SRL competences, through an integrated assessment approach (functional, educational, neurocognitive, and neuroimaging).

DETAILED DESCRIPTION:
Participants

30 children with CP, age-range between 8 and 15 years (elementary and middle school - 3rd grade to 9th grade), without cognitive impairments, will be selected. Agreements in partaking in the study are already in place with CP rehabilitation centers on the north of Portugal. Participants have already been evaluated through cognitive and neuropsychological tools. Specifically, children should present a cognitive performance at least in Medium- Low level (WISC-III) and should have eventual epilepsy episodes under control. Participants need to be able to use a computer and have internet access, and are required to have a native level of writing and reading skills in the Portuguese language.

Recruitment and selection

Recruitment will take place in the Portuguese associations of cerebral palsy. A collaboration agreement was established with the Federation of Portuguese Cerebral Palsy Associations (FPCPA), which includes 15 Cerebral Palsy Associations in Portugal. The Associations will evaluate their children and identify those who fulfil the inclusion criteria. The first contact with the parents/caregivers will be made by the associations and only after they accept to participate will the research team contact them. When identified, children and their parents will be debriefed, the consents delivered, explained, and signed.

Procedure

The FCPA (Federation Associations of Cerebral Palsy) will identified the needs to promote self-regulation skills and school involvement of children with CP. Researchers will established contact and held formal meetings with therapists to identify key difficulties and needs.

a) Two questions guided the meetings:

i. "What are the main difficulties you have while intervening with children with CP?" ii. "What do you think we could help with?" For study 4 a randomized controlled trial will be developed with three groups. After obtaining informed consent from parents/caregivers, participants meeting criteria will be randomly assigned to one condition. The control group (CG) will not have access to the online platform, i.e. no intervention. The intervention group 1 (IG1) will receive on a weekly basis tasks and activities on the online platform to promote SR and SE, as well as chapters of the narrative. The intervention group 2 (IG2) will receive the same tasks and materials as IG1 but embedded with Gamification Strategies.

Phase 1 - Selection of Gamification Strategies

Reeves and Read (2009) identify the "Ten Ingredients of Great Games" as good examples of elements of Gamification: i) self-representation with avatars, ii) three-dimensional environments, iii) narrative context, iv) feedback, v) reputations, ranks and levels, vi) marketplaces and economies, vii) competition under rules that are explicit and enforced, viii) teams, ix) parallel communication systems that can be easily configured, x) time pressure. Specifically, in the school context, a number of game elements have been identified as promoters of SE, contributing to learning success of students: collaboration and competition, feedback and reputations, ranks and levels, and reinforcement. Accordingly, through Canvas® Platform tools, these elements will be applied to the IG2. The project will be presented to FCPA, who will be involved in all stages.

Phase 2 - Implementation

The project will be presented at the rehabilitation centers, to technicians and parents/caregivers; and to children who accept to participate. The intervention will take place at the rehabilitation centers, and the collaboration of all stakeholders is imperative. Parents/caregivers will be asked to stimulate their child to engage with, and talk about, the intervention, and to contact the research team whenever is necessary. Secondly, parents/caregivers and children will fill-in the informed consents and the socio-demographic questionnaires. Each child will have a login through e-mail into the platform.

This intervention will take place during the weekly occupational therapy (OT) sessions at the rehabilitation centers to guarantee implementation of the research protocol (e.g., internet access).

Phase 3 - Program evaluation

To capture the procedural dimension of the phenomenon and evaluate the impact of the intervention on the promotion of SE, SRL, and EF in children with CP, several elements will be considered: aptitude (i.e. questionnaires), event (i.e. checklist, observations), and neuroplasticity, as suggested by the literature of SRL processes (Núñez, Rosário, Vallejo & González-Pienda, 2013; Zimmerman, 2008). The hypothesis is that the intervention will promote statistically significant improvements in the IG1 and IG2 in all measures - SE, SRL, EF evaluation, compared to the CG.

The evaluation protocol described refers to assessment that will be conducted with the children participating in the study. Children were assessed on their intellectual ability using the Wechsler Intelligence Scale for Children - Third Edition (WISC-III) (Wechsler, 2003). Medical and therapists' records were reviewed to collect information about the topographic motor type and quality of tonus, as well as the child's level on the Gross Motor Function Classification System (GMFCS) (Andrada, 2012; Palisano et al., 2015). Other variables were gathered: gender, date of birth, school grades from the last year, types of therapies each child is attending, extracurricular activities, internet access at home, computer access, story reading frequency, curricular adaptations.

The following measures will be collected before the start of the intervention, at the end, and 3 months after the intervention completion.

1. Neuropsychological assessment

   1. This investigation follows the Miyake model of EF. This model postulates that EF is comprised of three latent variables with different roles (Inhibition, Shifting, and Updating) that can be learned through the individual's performance (Miyake, Emerson, & Palisano et al., 2015). The CANTAB application was selected for the pre- post assessment. From the set of the CANTAB, 6 tests were selected: i. Multitasking Test (MTT) - To manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task- irrelevant information (Shifting).

   ii. One Touch Stockings of Cambridge (OTS) - To assess both the spatial planning and the working memory subdomains (Updating/Planning). Based upon the Tower of Hanoi test.

   iii. Stop Signal Task (SST) - To measure response inhibition and impulse control (Inhibition Control).

   iv. Spatial Working Memory (SWM) - To provide a measure of strategy and of working memory errors.

   v. Motor Screening Task (MOT) - To provide a general assessment of whether sensorimotor deficits or lack of comprehension will limit the collection of valid data from the participant.

   vi. Emotion Recognition Task (ERT) - This task, measures the ability to identify six basic emotions in facial expressions along a continuum of expression magnitude.

   b) Functional magnetic resonance imaging (FMRI)

   i. A classic test of inhibitory control (Go-No-go task) will be used; another test will be adapted using images from the e-book of the "Incredible Adventures of the Anastácio, the Explorer". 2. Self-Report Questionnaires

3. Effort Measures 4. Interviews

a) Self-Regulation Learning (Rosário et al., 2011)

i. SRL Strategies Inventory

1. Comprises nine self-regulated learning strategies presented in a Likert-like format of 5 points (1=never to 5=always)
2. Items assess the three phases of SRL model: PLEE (three items per each phase) i. Planning (e.g., ''I make a plan before I begin writing. I think about what I want to say and how I need to write it.'' - α=.80), ii. Execution (e.g., ''If I become distracted or lose concentration while I am in class or studying, then I usually try to regain my goals.'' - α=.85) iii. Evaluation (e.g., ''I compare the grades I receive with the goals I set for that subject.''- α=.87)

   b) Engagement

ii. School Engagement Scale (Fredricks et al., 2005)

1. The scale comprises 14 items presented in a Likert-like format of 5 points (1=never to 5=always).
2. Items cluster in the three SE dimensions (i.e., behavioral, emotional, and cognitive).

   i. Behavioral Engagement scale comprises 5 items (e.g., "I follow the rules at school.") (α=.77);

   ii. Emotional Engagement scale comprises 6 items (e.g., "I feel happy in school.) (α=.86); iii. Cognitive Engagement scale comprises 8 items (e.g., I study at home even when I don't have a test.) (α=.82).
   1. Throughout the interventions, children will be asked to complete different tasks on a voluntary basis (e.g., viewing videos, participation in the discussion forums).
   2. The fulfillment of these tasks and of the session's goals will be on-task measures of children's involvement with the intervention program

   <!-- -->

   1. Children, therapists, and parents/caregivers will be selected for a purposeful sample upon completion of the program.
   2. Interviews will be semi-structured to further understand the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children should present a cognitive performance at least in Medium- Low level (WISC-III);
* Children should have eventual epilepsy episodes under control;
* Participants need to be able to use a computer and have internet access, and are required to have a native level of writing and reading skills in the Portuguese language.

Exclusion Criteria:

-

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Neuropsychological assessment (CANTAB) - Executive function performance | pre (week 1) and post (up to 6 weeks) intervention
  This investigation follows the Miyake model of EF. This model postulates that EF is comprised of three latent variables, Inhibition, Shifting, and Updating, that can be learned through the individual's performance. The CANTAB application was selected to evaluate the baseline performance of the participant's pre-intervention and to evaluate the change in participant's performance after the intervention program, i.e., post-assessment. 6 tests were selected: Multitasking Test (Shifting); One Touch Stockings of Cambridge (Updating/Planning) - based upon the Tower of Hanoi test; Stop Signal Task (Inhibition Control); Spatial Working Memory - Working memory); Motor Screening Task (general assessment of sensorimotor deficits or lack of comprehension); Emotion Recognition Task (measure the ability to identify 6 basic emotions in facial expressions).
Functional magnetic resonance imaging (FMRI) | pre (week 1) and post (up to 6 weeks) intervention
  A classic test of inhibitory control (Go-No-go task) will be used; another test will be adapted using images from the e-book of the "Incredible Adventures of the Anastácio, the Explorer".
  The purpose of this two moments evaluation is assess the change in self-control performance and the impact in the neurocognitive structures and neural connections.
Self-Regulation Learning | pre (week 1) and post (up to 6 weeks) intervention
  SRL Strategies Inventory (Rosário et al., 2011)
  1. Comprises nine self-regulated learning strategies presented in a Likert-like format of 5 points (1=never to 5=always);
  2. Items assess the three phases of SRL model: PLEE (three items per each phase); i. Planning (e.g., ''I make a plan before I begin writing. I think about what I want to say and how I need to write it.'' - α=.80), ii. Execution (e.g., ''If I become distracted or lose concentration while I am in class or studying, then I usually try to regain my goals.'' - α=.85) iii. Evaluation (e.g., ''I compare the grades I receive with the goals I set for that subject.''- α=.87).
  A higher score in the SRL Strategies Inventory translates a better SRL perceived performance.
Engagement | pre (week 1) and post (up to 6 weeks) intervention
  School Engagement Scale (Fredricks et al., 2005)
  1. The scale comprises 14 items presented in a Likert-like format of 5 points (1=never to 5=always).
  2. Items cluster in the three SE dimensions (i.e., behavioral, emotional, and cognitive).
     i. Behavioral Engagement scale comprises 5 items (e.g., "I follow the rules at school.") (α=.77); ii. Emotional Engagement scale comprises 6 items (e.g., "I feel happy in school.) (α=.86); iii. Cognitive Engagement scale comprises 8 items (e.g., I study at home even when I don't have a test.) (α=.82).
     A higher score in the School Engagement Scale translates a better-perceived engagement with school.
Children Interviews | post intervention (up to 6 weeks)
  perceived intervention impact interview

SECONDARY OUTCOMES:
Effort Measures - platform records | daily basis (during 6 weeks)
  1. Throughout the interventions, children will be asked to complete different tasks on a voluntary basis (e.g., viewing videos, participation in the discussion forums).
  2. The fulfillment of these tasks and of the session's goals will be on-task measures of children's involvement with the intervention program.
Session Evaluation | weekly (during 6 weeks)
  The research team will develop a satisfaction questionnaire based on previous satisfaction instruments used with this population in a previous study with The Incredible Anastacio's Adventure (Pereira et al, 2019). The questionnaire will address aspects of utility and feasibility of the program and perceived support by the educational psychologist from the students' perspective.
  The questionnaire comprises 23 items with a 5 point Likert scale (1=never to 5=always).
  A higher score in the Satisfaction questionnaire translates a better-perceived satisfaction with the intervention program.

CONTACTS AND LOCATIONS:
Locations (1):
- Associação Paralisia Cerebral, Braga, Portugal

REFERENCES:
- See also: Description Research group website — http://www.guia-psi.com/paralisia-cerebral.html